CLINICAL TRIAL: NCT04307550
Title: Inhaled Isopropyl Alcohol Versus Placebo to Manage Nausea at Electronic Dance Music Festivals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony Seto (Other)
Responsible Party: Sponsor-Investigator, Anthony Seto, Course Chair, "Intro to Clinical Practice", University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB20-0288
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — 2-Propanol; Ethanol; Protein-Arginine Deiminases

STUDY DESIGN:
Intervention Model Description: Participants in Arm 1 will nasally inhale an isopropyl alcohol pad with 10 inhalations (intervention). Participants in Arm 2 will nasally inhale a sterile saline pad of similar appearance with 10 inhalations (placebo).
Who Masked: Participant, Outcomes Assessor
Masking Description: An intervention/care provider will remove the packaging so that participants will be unable to identify the inhaled substance. We acknowledge that the smell of isopropyl alcohol may be familiar and thus identifiable for some treatment arm participants. However, participants will not be informed of the identity of the treatment and placebo during the consent process, instead only being told that we are comparing two inhaled substances to assess their relative effectiveness. Thus, recognizing they are inhaling isopropyl alcohol should not bias participants' responses, given they will not know whether isopropyl alcohol is a treatment or control.
  The outcomes assessor will be blinded, because the randomization and intervention delivery are both completed by the intervention/care provider, who will not be involved in screening/baseline assessment nor outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isopropyl Alcohol (Experimental): 10 inhalations of an isopropyl alcohol pad held within 2cm from the nares
  Interventions: Drug: Isopropyl alcohol
- Sterile Saline (Placebo Comparator): 10 inhalations of a sterile saline pad held within 2cm from the nares
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Isopropyl alcohol — 10 inhalations of an isopropyl alcohol pad
  Other Names: Isopropyl alcohol pad
  Arms: Isopropyl Alcohol
Other: Placebo — 10 inhalations of a sterile saline pad
  Other Names: Sterile saline pad
  Arms: Sterile Saline

SUMMARY:
BACKGROUND

Studies have shown that isopropyl alcohol inhalation is effective for the relief of nausea in the emergency department. A 2016 randomized controlled trial found that nasally inhaled isopropyl alcohol achieved better nausea relief compared to placebo during a 10-minute period. In 2018, another randomized controlled trial showed that nasally inhaled isopropyl alcohol with or without oral ondansetron provided greater relief for nausea than oral ondansetron alone.

QUESTION

In electronic dance music festival attendees, who present with nausea to the medical team, how does inhaled isopropyl alcohol compare with inhaled sterile saline (placebo) for self-reported nausea 10-minutes post-intervention?

METHODS

Canadian electronic dance music festival attendees who present with nausea to the medical team, will be recruited until sample size reaches at least 70. Inclusion criteria will be festival attendees aged 18+ with a complaint of nausea. Exclusion criteria will include known allergy to isopropyl alcohol, inability to inhale through the nares, inability to report level of nausea, or already have taken an anti-nauseant.

After obtaining consent, participants will be randomized into two study arms. Arm 1 will nasally inhale an isopropyl alcohol pad with 10 deep inhalations (intervention). Arm 2 will nasally inhale a sterile saline pad with 10 deep inhalations (placebo). The pad must be within 2cm from the nares to ensure delivery. According to a study in 2002, isopropyl alcohol pad inhalation, dosed at 3 inhalations every 5 minutes for 3 doses, was not significantly different than standard treatment for relief of nausea. 10 inhalations exceeds the 9-dose total reported in the paper, and a one-time bolus dose of 10 inhalations, for the population and festival context, is more feasible in terms of patient compliance and patient flow.

After randomization, participants will rate their nausea on a numeric response scale (0 to 10, where 0 is no nausea and 10 is "worst nausea imaginable"). 10-minutes post-inhalation (isopropyl alcohol or placebo), participants will be asked to rate their nausea again.

The primary outcome is self-reported nausea scores 10-minutes post-intervention. The secondary outcome is the presence or absence of any vomiting spells 10-minutes post-intervention, as well as the presence or absence of rescue-medication needed 10-minutes post-intervention.

DETAILED DESCRIPTION:
POPULATION OF INTEREST

Participants will be recruited from electronic dance music (EDM) festivals in Canada. This population was chosen because festival participants often present to event medical staff with a complaint of nausea, in a setting where the availability of medical resources such as oral and intravenous anti-nauseants are more limited than an emergency department. Although the effectiveness of isopropyl alcohol pads as anti-nauseant therapy has been demonstrated in hospital emergency rooms, no prior studies, to the investigators' knowledge, have assessed outcomes in festival populations. This study will be conducted by adapting protocols from prior studies that examined the effects of inhaled isopropyl alcohol on patient-reported nausea and will add to the current state of knowledge by investigating a novel population.

EDM events are included in this study, because the investigators have long-standing experience working at these festivals as part of the main medical team, responsible for providing medical care to all festival participants. Odyssey Medical, the organization that oversees all medical staff at these EDM events, has granted the investigators permission to integrate the proposed research study into patient care at these festivals. This organization recruits multi-disciplinary volunteers (physicians, nurses, respiratory therapists, pharmacists, lifeguards, paramedics, and first aiders) to manage the medical needs of festival attendees.

PARTICIPANT SCREENING

Participants will verbally respond to screening questions, with responses recorded electronically by Research Personnel #1 (aka "the assessor") on a secure Google Form (printed copies will be available as back-up). Individuals who satisfy all inclusion/exclusion criteria will continue in the study, while those who do not meet criteria will receive standard medical care as needed (e.g. oral or intravenous anti-nauseant).

Consent to participate in the study will be obtained with a signature, after review of a written consent form. For the consent process, the investigators will have a witness from the medical team. For all individuals with a complaint of nausea, the assessor will outline the purpose of the study, clarify risks/benefits, and highlight that participation is voluntary and can be withdrawn, before seeking consent. Given that festival participants may be intoxicated with substances, Research Personnel #1 will determine whether the participant has the mental capacity to continue with the study. Research Personnel #1 will confirm the person's name, sex, and age. If the participant is unable to report their name, sex, and age accurately (using the patient's chart as a comparator or a friend/family member), then this implies that the participant is not oriented enough (e.g., potentially too intoxicated) to continue the study; this participant would not continue with the study. Also, if the participant cannot verbalize a pre-treatment nausea score (e.g., tries to communicate with fingers or body language, asks a friend to translate, etc.), then this implies that they may be too intoxicated to use their own cognitive capacity to determine a specific number and then verbalize it; this participant would not continue with the study.

If consent is granted, the following information about the participant will be collected throughout the study:

* Numerical identification number (will be assigned based on the order of recruitment, e.g. participant 001, participant 002)
* Age
* Sex
* Self-reported alcohol consumed
* Self-reported recreational drugs ingested
* Self-reported other suspected contributors of nausea (e.g. migraine, head injury, pregnancy, infection)
* Pre-treatment nausea level (0-11)
* Absence/presence of emesis prior to treatment
* 10-minute post-treatment nausea level (0-11)
* Absence/presence of emesis post-treatment
* Any side effects or additional symptoms post-treatment

No uniquely identifying information such as name, birth date, or Provincial Health Care number will be recorded at any point of the study to preserve anonymity. Age and sex will be recorded alongside screening criteria and will be linked with each individual's data for future subgroup analyses, but this broad information is not expected to interfere with anonymity.

PARTICIPANT RANDOMIZATION

Included participants will be assigned to one of two study arms through randomization, facilitated by an electronic random number generator operated by Research Personnel #2 (i.e. "the intervention provider"), who will not be present for the baseline screening assessment.

INTERVENTION DELIVERY

Research Personnel #2 will then deliver the intervention according to the assigned study arm. Participants in Arm 1 will nasally inhale an isopropyl alcohol pad with 10 inhalations (intervention). Participants in Arm 2 will nasally inhale a sterile saline pad of similar appearance with 10 inhalations (placebo). Research Personnel #2 will remove the packaging out of participants' sight, in order to ensure participants are blinded to the identity of the inhaled substance. The isopropyl alcohol pad, or sterile saline pad, will be held within 2cm of participants' nares to ensure delivery during inhalations, as a 2018 study demonstrated success using isopropyl alcohol aromatherapy as an anti-nauseant when inhaled from 1-2cm from the nares.

According to a 2002 study, isopropyl alcohol pad inhalation, dosed at 3 inhalations every 5 minutes for 3 doses, was not significantly different than standard anti-nauseant treatment for relief of nausea. 10 inhalations exceeds the 9-dose total reported in the paper, and a one time bolus dose of 10 inhalations, for this population and festival context, is more feasible in terms of patient compliance and patient flow in the main medical area. Two other studies' protocols involved inhaling isopropyl alcohol, as many times as participants desired, within a few minutes. With all protocols taken into consideration, the investigators have determined that 10 inhalations is an appropriate threshold for potential anti-nauseant effect.

OUTCOME ASSESSMENT

After Research Personnel #2 (aka "the intervention provider") has ensured that the intervention/placebo has been inhaled, they will leave the participant's bedside to prevent them from biasing any subsequent outcome assessment, given their knowledge of the study arm. The intervention provider will not disclose the identity of the inhaled substance to the participant nor to the assessor.

10 minutes post-inhalation, Research Personnel #1 (aka "the assessor"), will return and assess the participant's nausea using the same 11-point numerical scale prior to treatment. Participants will also be asked to report any new symptoms in order to aid the identification of possible adverse outcomes. Presence or absence of vomiting pre- and post-intervention will also be recorded.

After the data collection is complete, both the intervention and control arms will be offered further treatment by medical staff if their nausea has not subsided. These "rescue" (additional) therapies may include oral and/or intravenous anti-nauseants. The need for rescue medications will be recorded.

DATA ANALYSIS

For primary and secondary outcomes, data will be analyzed with a one-tailed repeated-measures t-test to see if there are any differences in self-reported nausea pre-intervention and 10-minutes post-intervention, between the means of the treatment arms.

Subgroup analyses will be performed, via repeated-measures t-test to see if there are any differences between the means of the treatment arms, by male sex, female sex, age (18-25, 25-34, 35+), alcohol ingested, any recreational substance ingested, alcohol plus other any recreational substance ingested, and self-reported other suspected contributors of nausea.

SAMPLE SIZE

Sample size for each group was calculated with the assumption that the outcome data fits a ratio scale (nausea is rated on a continuum, ranging from 0 to 10).

A sample size, for adequate study power, was performed with the following parameters:

* Study group design: two independent study groups
* Primary endpoint: continuous (means)
* Anticipated mean for isopropyl alcohol swab group: 3 +/- 3
* Anticipated mean for placebo group: 5
* Alpha: 0.05
* Power: 0.8

Previous work in 2016 found the median nausea score for the isopropyl alcohol pad group was 3 and for the placebo group, 6, in the emergency department. The investigators lowered the placebo group by 1 point, to 5, to be conservative in calculations. A 2018 study found that the standard deviation was up to 30, on scale of 0 to 100, for all treatment groups (when comparing inhaled isopropyl alcohol + oral ondansetron, inhaled isopropyl alcohol + oral placebo, and inhaled placebo + oral ondansetron); therefore, the investigators assume a standard deviation of up to 3, in their scale from 0 to 10.

The investigators calculated a minimum sample size of 46 to power the study. Given that the sample size is large enough, the central limit theorem supports the normality assumption; therefore, a parametric test was selected (repeated-measures t-test) for statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Festival attendees aged 18+
* A complaint of nausea of at least 1 on a scale of 0 to 10 (11-point scale, where 0 represents "no nausea" and 10 represents "worst nausea imaginable").

Exclusion Criteria:

* Known allergy to isopropyl alcohol (standard practice involves medical team members asking patients what allergies they have; we will not directly ask about isopropyl alcohol in order to keep participants blinded to interventions)
* Inability to inhale through the nares (e.g. distorted nasal anatomy, active nosebleed, obstructed nasal passages, rhinitis, anosmia)
* Inability to verbally report level of nausea
* Prior administration of an oral or intravenous anti-nauseant (e.g. metoclopramide, ondansetron, dimenhydrinate) by festival medical staff since arrival at the festival (would confound treatment effect)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Self-reported nausea scores | 10-minutes post-intervention
  Nausea rated on an 11-point scale (0 = "no nausea", 10 = "worst nausea imaginable")

SECONDARY OUTCOMES:
Presence of vomiting | 10-minutes post-intervention
  Presence (1) or absence (0) of any vomiting spells
Use of rescue-medication (i.e. oral/intravenous anti-nauseant) | 10-minutes post-intervention
  Presence (1) or absence (0) of any rescue-medication (i.e. oral/intravenous anti-nauseant), identified by patient's chart

CONTACTS AND LOCATIONS:
Overall Officials: Anthony V Seto, MD, Principal Investigator — University of Calgary
Locations (9):
- Canada (9):
  - Badlands Music Festival, Calgary, Alberta
  - Chasing Summer Music Festival, Calgary, Alberta
  - Family Reunion Music Festival, Calgary, Alberta
  - Bomfest Music Festival, Edmonton, Alberta
  - Hard West Music Festival, Wimborne, Alberta
  - Electronic dance music festivals in Calgary, Calgary
  - Electronic dance music festivals in Edmonton, Edmonton
  - Electronic dance music festivals in Toronto, Toronto
  - Electronic dance music festivals in Vancouver, Vancouver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] April MD, Oliver JJ, Davis WT, Ong D, Simon EM, Ng PC, Hunter CJ. Aromatherapy Versus Oral Ondansetron for Antiemetic Therapy Among Adult Emergency Department Patients: A Randomized Controlled Trial. Ann Emerg Med. 2018 Aug;72(2):184-193. doi: 10.1016/j.annemergmed.2018.01.016. Epub 2018 Feb 17. PMID 29463461
- [Background] Beadle KL, Helbling AR, Love SL, April MD, Hunter CJ. Isopropyl Alcohol Nasal Inhalation for Nausea in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2016 Jul;68(1):1-9.e1. doi: 10.1016/j.annemergmed.2015.09.031. Epub 2015 Dec 8. PMID 26679977
- [Background] Merritt BA, Okyere CP, Jasinski DM. Isopropyl alcohol inhalation: alternative treatment of postoperative nausea and vomiting. Nurs Res. 2002 Mar-Apr;51(2):125-8. doi: 10.1097/00006199-200203000-00009. PMID 11984383